CLINICAL TRIAL: NCT02423486
Title: The Comparison of Efficacy Between Electromagnetic Stimulation Therapy and Electromagnetic Stimulation Therapy With Extracorporeal Biofeedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-11-088; ksleedr (Other: Samsung Medical Center)
Record Dates: First submitted 2015-03-24; First posted 2015-04-22 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Urinary Stress Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Biofeedback, Psychology

ARMS (2):
- Electromagnetic stimulation therapy (Experimental): Electromagnetic stimulation therapy group
  Interventions: Device: Electromagnetic stimulation therapy (BIOCON-2000)
- Electromagnetic stimulation therapy with biofeedback (Experimental): Electromagnetic stimulation therapy with biofeedback group
  Interventions: Device: Electromagnetic stimulation therapy with biofeedback

INTERVENTIONS:
Device: Electromagnetic stimulation therapy (BIOCON-2000)
  Arms: Electromagnetic stimulation therapy
Device: Electromagnetic stimulation therapy with biofeedback
  Arms: Electromagnetic stimulation therapy with biofeedback

SUMMARY:
The aim of this study is to compare the efficacy between Electromagnetic Stimulation therapy and Electromagnetic Stimulation therapy with Extracorporeal Biofeedback in Stress Urinary Incontinence patient.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient with Stress Urinary Incontinence, over 20
2. Leakage over 2g in stress pad test
3. Capable of understanding and having signed the informed consent form after full discussion of the research nature of the treatment and its risks and benefits

Exclusion Criteria:

1. Mixed Urinary Incontinence which is dominant in urge urinary incontinence.
2. True incontinence
3. Overflow incontinence
4. Patient who had performed electric stimulation therapy,bladder training within 2 weeks before baseline.
5. Urinary tract infection found In urine test.
6. Patient who had pelvic organ prolapse.
7. Patient who had inserted pacemaker.
8. Pregnant woman, patient who have positive result in urine pregnancy test, patient who have plan pregnancy during study period.
9. Disorder in Neurosystem like stroke, multiple sclerosis, spinal injury, Parkinson's disease .
10. Patient who will participate in other clinical trial during this study.
11. Any other condition which, in the opinion of the investigator, makes the patient unsuitable for inclusion

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-11; Primary Completion 2019-09-06 (Actual); Study Completion 2019-11-28 (Actual)

PRIMARY OUTCOMES:
Rate comparison of complete recovery in stress pad test after 12 weeks of treatment | 12 weeks
  Complete recovery is defined as urinary leakage below than 2 gram in stress pad test.

SECONDARY OUTCOMES:
Incontinence Severity VAS at baseline,4weeks,8weeks,12weeks after treatment | 12 weeks
Sandvik questionnaire at baseline,4weeks,8weeks,12weeks after treatment | 12 weeks
Incontinence - Quality of Life questionnaire at baseline,8weeks,12 weeks after treatment | 12 weeks
Benefit,Satisfaction and Willingness to Continue questionnaire at 12 weeks after treatment | 12 weeks
Pelvic floor muscular strength at baseline,4weeks,8weeks,12weeks after treatment | 12 weeks
  Intravaginal pressure, Extracorporeal pelvic floor muscular strength, Oxford Scale at baseline,4weeks,8weeks,12weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kyu-Sung Lee, Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea